CLINICAL TRIAL: NCT01203722
Title: Reduced Intensity, Partially HLA Mismatched Allogeneic BMT for Hematologic Malignancies Using Donors Other Than First-degree Relatives
Brief Title: Reduced Intensity, Partially HLA Mismatched BMT to Treat Hematologic Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1055; NA_00039823 (Other: JHM IRB); P01CA015396 (NIH)
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hematologic Malignancies
Keywords: Reduced intensity; partially HLA mismatched allogeneic BMT; Acute leukemias; Chronic leukemias; Myelodysplasia; Lymphomas; Unrelated or non-first-degree related donors; Peripheral blood stem cell transplant
MeSH Terms: conditions — Hematologic Neoplasms; Anemia, Refractory, with Excess of Blasts; Lymphoma | interventions — fludarabine; Cyclophosphamide; Whole-Body Irradiation; Peripheral Blood Stem Cell Transplantation; Mycophenolic Acid; Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- REGIMEN B (Active Comparator): Pre-BMT :
  * Day -6 through -2: Fludarabine 30 mg/m2/day (adjusted for renal function; maximum cumulative dose, 150 mg/m2) administered IV
  * Day -6 and -5: Cytoxan 14.5 mg/kg/day administered IV
  * Day -1: 400 cGy total body irradiation (TBI) administered in a single fraction
  Day 0: Allogeneic blood or marrow transplantation (BMT)
  Post-Transplantation Immunosuppression Consisting of:
  * Day 3 and 4: High-dose Cytoxan 50mg/kg/day (adjusted according to IBW) administered IV
  * Day 5: Sirolimus loading dose 6 mg PO once
  * Day 5 thru Day 35: Mycophenolate Mofetil (MMF) 15 mg/kg PO TID (maximum daily dose 3 g/day)
  * Day 6 thru Day 180: Sirolimus maintenance dose 2 mg PO QD with dose adjustments to maintain trough of 3 - 12 ng/mL
  Interventions: Drug: Fludarabine; Drug: Cytoxan; Radiation: Total Body Irradiation; Procedure: Allogeneic Blood or Marrow Transplant; Drug: Mycophenolate Mofetil; Drug: Sirolimus
- REGIMEN C (Active Comparator): Pre-BMT:
  * Day -6 through -2: Fludarabine 30 mg/m2/day (adjusted for renal function; maximum cumulative dose, 150 mg/m2) administered IV
  * Day -6 and -5: Cytoxan 14.5 mg/kg/day administered IV
  * Day -1: 400 cGy TBI administered in a single fraction
  Day 0: BMT
  Post-Transplantation Immunosuppression Consisting of:
  * Day 3 and 4: High-dose Cytoxan 50mg/kg/day (adjusted according to IBW) administered IV
  * Day 5 thru Day 35: MMF 15 mg/kg PO TID (maximum daily dose 3 g/day)
  * Day 5 thru Day 180: Tacrolimus 1 mg administered IV QD
  Interventions: Drug: Fludarabine; Drug: Cytoxan; Radiation: Total Body Irradiation; Procedure: Allogeneic Blood or Marrow Transplant; Drug: Mycophenolate Mofetil; Drug: Tacrolimus
- REGIMEN B2 (Active Comparator): Pre-PBSCT:
  * Day -6 through -2: Fludarabine 30 mg/m2/day (adjusted for renal function; maximum cumulative dose, 150 mg/m2) administered IV
  * Day -6 and -5: Cytoxan 14.5 mg/kg/day administered IV
  * Day -1: 400 cGy TBI administered in a single fraction
  Day 0: Peripheral Blood Stem Cell Transplant (PBSCT)
  Post-Transplantation Immunosuppression Consisting of:
  * Day 3 and 4: High-dose Cytoxan 50mg/kg/day (adjusted according to IBW) administered IV
  * Day 5: Sirolimus loading dose 6 mg PO once
  * Day 5 thru Day 35: MMF 15 mg/kg PO TID (maximum daily dose 3 g/day)
  * Day 6 thru Day 180: Sirolimus maintenance dose 2 mg PO QD with dose adjustments to maintain trough of 3 - 12 ng/mL
  Interventions: Drug: Fludarabine; Drug: Cytoxan; Radiation: Total Body Irradiation; Procedure: Peripheral Blood Stem Cell Transplant; Drug: Mycophenolate Mofetil; Drug: Sirolimus
- REGIMEN B3: HIV patients with CCRd32 homozygous donors (Active Comparator): Pre-PBSCT:
  * Day -6 through -2: Fludarabine 30 mg/m2/day (adjusted for renal function; maximum cumulative dose, 150 mg/m2) administered IV
  * Day -6 and -5: Cytoxan 14.5 mg/kg/day administered IV
  * Day -1: 400 cGy TBI administered in a single fraction
  Day 0: Peripheral Blood Stem Cell Transplant (PBSCT)
  Post-Transplantation Immunosuppression Consisting of:
  * Day 3 and 4: High-dose Cytoxan 50mg/kg/day (adjusted according to IBW) administered IV
  * Day 5: Sirolimus loading dose 6 mg PO once
  * Day 5 thru Day 35: MMF 15 mg/kg PO TID (maximum daily dose 3 g/day)
  * Day 6 thru Day 180: Sirolimus maintenance dose 2 mg PO QD with dose adjustments to maintain trough of 3 - 12 ng/mL
  Interventions: Drug: Fludarabine; Drug: Cytoxan; Radiation: Total Body Irradiation; Procedure: Peripheral Blood Stem Cell Transplant; Drug: Mycophenolate Mofetil; Drug: Sirolimus

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 30 mg/m2/day
Drug: Cytoxan — Pre-BMT: Cytoxan 14.5 mg/kg/day administered IV; Post-Transplantation: High-dose Cytoxan 50mg/kg/day
  Other Names: High-dose Cytoxan
Radiation: Total Body Irradiation — 400 cGy TBI administered in a single fraction
  Other Names: TBI
Procedure: Allogeneic Blood or Marrow Transplant
  Other Names: BMT
  Arms: REGIMEN B; REGIMEN C
Procedure: Peripheral Blood Stem Cell Transplant
  Other Names: PBSCT
  Arms: REGIMEN B2; REGIMEN B3: HIV patients with CCRd32 homozygous donors
Drug: Mycophenolate Mofetil — 15mg/kg by mouth three times daily
  Other Names: MMF
Drug: Sirolimus — Loading Dose: Sirolimus 6mg by mouth once; Maintenance dose: Sirolimus 2mg by mouth daily
  Arms: REGIMEN B; REGIMEN B2; REGIMEN B3: HIV patients with CCRd32 homozygous donors
Drug: Tacrolimus — Tacrolimus 1mg intravenously, daily
  Arms: REGIMEN C

SUMMARY:
If transplantation using mismatched unrelated donors or non-first-degree relatives could be performed with an acceptable toxicity profile, an important unmet need would be served. Towards this goal, the current study extends our platform of nonmyeloablative, partially HLA-mismatched bone marrow transplant (BMT) and Peripheral Blood Stem Cell Transplant (PBSCT) to the use of such donors, investigating up to several postgrafting immunosuppression regimens that incorporate high-dose Cy. Of central interest is the incorporation of sirolimus into this postgrafting immunosuppression regimen.

The primary goal for phase 1 is to identify a transplant regimen associated with acceptable rates of severe acute GVHD and NRM by Day 100 and for phase 2 estimate the 6-month probability of survival without having had acute grade III- IV GVHD or graft failure.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Patient age 0.5-75 years
2. Absence of a suitable related or unrelated bone marrow donor who is molecularly matched at HLA-A, B, Cw, DRB1, and DQB1.
3. Absence of a suitable partially HLA-mismatched (haploidentical), first-degree related donor. Donors who are homozygous for the CCR5delta32 polymorphism are given preference.
4. Eligible diagnoses:

   1. Relapsed or refractory acute leukemia in second or subsequent remission, with remission defined as <5% bone marrow blasts morphologically
   2. Poor-risk acute leukemia in first remission, with remission defined as <5% bone marrow blasts morphologically:

      * AML with at least one of the following:

        * AML arising from MDS or a myeloproliferative disorder, or secondary AML
        * Presence of Flt3 internal tandem duplications
        * Poor-risk cytogenetics: Complex karyotype [> 3 abnormalities], inv(3), t(3;3), t(6;9), MLL rearrangement with the exception of t(9;11), or abnormalities of chromosome 5 or 7
        * Primary refractory disease
      * ALL (leukemia and/or lymphoma) with at least one of the following:

        * Adverse cytogenetics such as t(9;22), t(1;19), t(4;11), or MLL rearrangement
        * Clear evidence of hypodiploidy
        * Primary refractory disease
      * Biphenotypic leukemia
   3. MDS with at least one of the following poor-risk features:

      * Poor-risk cytogenetics (7/7q minus or complex cytogenetics)
      * IPSS score of INT-2 or greater
      * Treatment-related MDS
      * MDS diagnosed before age 21 years
      * Progression on or lack of response to standard DNA-methyltransferase inhibitor therapy
      * Life-threatening cytopenias, including those generally requiring greater than weekly transfusions
   4. Interferon- or imatinib-refractory CML in first chronic phase, or non-blast crisis CML beyond first chronic phase.
   5. Philadelphia chromosome negative myeloproliferative disease.
   6. Chronic myelomonocytic leukemia.
   7. Juvenile myelomonocytic leukemia.
   8. Low-grade non-Hodgkin lymphoma (including SLL and CLL) or plasma cell neoplasm that has:

      * progressed after at least two prior therapies (excluding single agent rituximab and single agent steroids), or
      * in the case of lymphoma undergone histologic conversion;
      * patients with transformed lymphomas must have stable disease or better.
   9. Poor-risk CLL or SLL as follows:

      * 11q deletion disease that has progressed after a combination chemotherapy regimen,
      * 17p deletion disease,
      * or histologic conversion;
      * patients with transformed lymphomas must have stable disease or better.
   10. Aggressive non-Hodgkin lymphoma as follows, provided there is stable disease or better to last therapy:

       * NK or NK-T cell lymphoma, hepatosplenic T-cell lymphoma, or subcutaneous panniculitic T-cell lymphoma, blastic/ blastoid variant of mantle cell lymphoma
       * Hodgkin or aggressive non Hodgkin lymphoma that has failed at least one multiagent regimen, and the patient is either ineligible for autologous BMT or autologous BMT is not recommended.
       * Eligible subtypes of aggressive non-Hodgkin lymphoma include:

         * mantle cell lymphoma
         * follicular grade 3 lymphoma
         * diffuse large B-cell lymphoma or its subtypes, excluding primary CNS lymphoma
         * primary mediastinal large B-cell lymphoma
         * large B-cell lymphoma, unspecified
         * anaplastic large cell lymphoma, excluding skin-only disease
         * Burkitt's lymphoma or atypical Burkitt's lymphoma (high-grade B-cell lymphoma, unclassifiable, with features intermediate between diffuse large B-cell lymphoma and Burkitt's), in complete remission
5. Patients with CLL, SLL, or prolymphocytic leukemia must have < 20% bone marrow involvement by malignancy (to lower risk of graft rejection).
6. One of the following, in order to lower risk of graft rejection:

   * Cytotoxic chemotherapy, an adequate course of 5-azacitidine or decitabine, or alemtuzumab within 3 months prior to start of conditioning; or
   * Previous BMT within 6 months prior to start of conditioning.

   NOTE: Patients who have received treatment outside of these windows may be eligible if it is deemed sufficient to reduce graft rejection risk; this will be decided on a case-by-case basis by the PI or co-PI.
7. Any previous BMT must have occurred at least 3 months prior to start of conditioning.
8. Adequate end-organ function as measured by:

   1. Left ventricular ejection fraction greater than or equal to 35%, or shortening fraction > 25%, unless cleared by a cardiologist
   2. Bilirubin ≤ 3.0 mg/dL (unless due to Gilbert's syndrome or hemolysis), and ALT and AST < 5 x ULN
   3. FEV1 and FVC > 40% of predicted; or in pediatric patients, if unable to perform pulmonary function tests due to young age, oxygen saturation >92% on room air
9. ECOG performance status < 2 or Karnofsky or Lansky score > 60

Patient Exclusion Criteria:

* Not pregnant or breast-feeding.
* No uncontrolled bacterial, viral, or fungal infection.

  * Note: HIV-infected patients are potentially eligible. Eligibility of HIV-infected patients will be determined on a case-by-case basis.
* No previous allogeneic BMT (syngeneic BMT permissible).
* Active extramedullary leukemia or known active CNS involvement by malignancy. Such disease treated into remission is permitted.

Donor Inclusion Criteria:

1. Potential donors consist of:

   * Unrelated donors
   * Second-degree relatives
   * First cousins
2. The donor and recipient must be identical at at least 5 HLA alleles based on high resolution typing of HLA-A, -B, -Cw, -DRB1, and -DQB1, with at least one allele matched for a HLA class I gene (HLA-A, -B, or -Cw) and at least one allele matched for a class II gene (HLA-DRB1 or -DQB1).
3. Meets institutional selection criteria and medically fit to donate. 4 . Lack of recipient anti-donor HLA antibody. Note: In some instances, low level, non-cytotoxic HLA specific antibodies may be permissible if they are found to be at a level well below that detectable by flow cytometry. This will be decided on a case-by-case basis by the PI and one of the immunogenetics directors. Pheresis to reduce anti-HLA antibodies is permissible; however eligibility to proceed with the transplant regimen would be contingent upon the result.

Donor Exclusion Criteria:

* Donor must not be HLA identical to the recipient.
* Has not donated blood products to recipient.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Transplant regimen as determined by rates of severe acute graft-versus-host-disease (GVHD) | Study Day 100
  Two immunosuppressive regimens with Fludarabine-Cytoxan-TBI conditioning will be studied in reduced-intensity, partially HLA mismatched allogeneic BMT from unrelated or non-first-degree related donors. Transplant regimen will be determined by acceptable rates of severe acute GVHD (< 25%).
Transplant regimen as determined by rates of transplant-related nonrelapse mortality (NRM) | Study Day 100
  Two immunosuppressive regimens with Fludarabine-Cytoxan-TBI conditioning will be studied in reduced-intensity, partially HLA mismatched allogeneic BMT from unrelated or non-first-degree related donors. Transplant regimen will be determined by acceptable rates transplant-related NRM (< 20%).
6-month probability of survival as assessed by absence of grade III-IV GVHD or evidence of graft failure. | 6 months
  Two immunosuppressive regimens with Fludarabine-Cytoxan-TBI conditioning will be studied in reduced-intensity, partially HLA mismatched allogeneic BMT from unrelated or non-first-degree related donors.

SECONDARY OUTCOMES:
Progression-free survival | 7 years
  All patients will be tracked from Day 0 to date of first objective disease progression, death from any cause, or last patient evaluation. Patients who have not progressed or died will be censored at the last date they were assessed and deemed free of relapse or progression.
Event-free survival | 7 years
  All patients will be tracked from Day 0 to date of first objective disease progression, death from any cause, or last patient evaluation. Patients who have not progressed or died will be censored at the last date they were assessed and deemed free of relapse or progression.
Overall survival | 7 years
  All patients will be tracked from Day 0 to date of first objective disease progression, death from any cause, or last patient evaluation. Patients who have not progressed or died will be censored at the last date they were assessed and deemed free of relapse or progression.
Cumulative incidence of progression or relapse | 7 years
  All patients will be tracked from Day 0 to date of first objective disease progression, death from any cause, or last patient evaluation. Patients who have not progressed or died will be censored at the last date they were assessed and deemed free of relapse or progression.
Cumulative incidence of NRM. | 7 years
  All patients will be tracked from Day 0 to date of first objective disease progression, death from any cause, or last patient evaluation. Patients who have not progressed or died will be censored at the last date they were assessed and deemed free of relapse or progression.
Cumulative incidence of acute grade II-IV GVHD. | 1 year
  All suspected cases of acute GVHD must be confirmed histologically by biopsy of an affected organ (skin, liver, or gastrointestinal tract). Date of symptom onset, date of biopsy confirmation of GVHD, maximum clinical grade, and dates and types of treatment will be recorded. Dates of symptom onset of grade II or higher GVHD and grade III-IV GVHD will be recorded.
Cumulative incidence of acute grade III-IV GVHD | 1 year
  All suspected cases of acute GVHD must be confirmed histologically by biopsy of an affected organ (skin, liver, or gastrointestinal tract). Date of symptom onset, date of biopsy confirmation of GVHD, maximum clinical grade, and dates and types of treatment will be recorded. Dates of symptom onset of grade II or higher GVHD and grade III-IV GVHD will be recorded.
Cumulative incidence of chronic GVHD | 1 year
  All suspected cases of acute GVHD must be confirmed histologically by biopsy of an affected organ (skin, liver, or gastrointestinal tract). Date of symptom onset, date of biopsy confirmation of GVHD, maximum clinical grade, and dates and types of treatment will be recorded. Dates of symptom onset of grade II or higher GVHD and grade III-IV GVHD will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ambinder, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Rappazzo KC, Zahurak M, Bettinotti M, Ali SA, Ambinder AJ, Bolanos-Meade J, Borrello I, Dezern AE, Gladstone D, Gocke C, Fuchs E, Huff CA, Imus PH, Jain T, Luznik L, Rahmat L, Swinnen LJ, Wagner-Johnston N, Jones RJ, Ambinder RF. Nonmyeloablative, HLA-Mismatched Unrelated Peripheral Blood Transplantation with High-Dose Post-Transplantation Cyclophosphamide. Transplant Cell Ther. 2021 Nov;27(11):909.e1-909.e6. doi: 10.1016/j.jtct.2021.08.013. Epub 2021 Aug 20. PMID 34425261
- [Derived] Kasamon YL, Ambinder RF, Fuchs EJ, Zahurak M, Rosner GL, Bolanos-Meade J, Levis MJ, Gladstone DE, Huff CA, Swinnen LJ, Matsui WH, Borrello I, Brodsky RA, Jones RJ, Luznik L. Prospective study of nonmyeloablative, HLA-mismatched unrelated BMT with high-dose posttransplantation cyclophosphamide. Blood Adv. 2017;1(4):288-292. doi: 10.1182/bloodadvances.2016002766. Epub 2017 Jan 6. PMID 29242852

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT01203722/Prot_SAP_001.pdf